CLINICAL TRIAL: NCT05116696
Title: Comparison of Short- and Long Term Clinical Outcomes of Patients With Stage IV Chronic Limb-threatening Ischemia and Colorectal Cancer Liver Metastases
Brief Title: Comparison of Outcomes of Patients With Stage IV Chronic Limb-threatening Ischemia and Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Petar Zlatanovic, Principal Investigator, Clinical Centre of Serbia
Other Study IDs: CltiCancer
Record Dates: First submitted 2021-10-27; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Chronic Limb-Threatening Ischemia; Colorectal Carcinoma; Colorectal Carcinoma Metastatic in the Liver
Keywords: Peripheral Arterial Disease (PAD); Chronic Limb-Threatening Ischemia (CLTI); Colorectal Carcinoma (CRC); Colorectal Liver Metastases (CRLM)
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Colorectal Neoplasms; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic limb-threatening ischemia (CLTI) group: All CLTI patients presenting with wound, ischemia, foot infection (WIfI) stage IV disease consecutively treated at one institution
  Interventions: Procedure: For chronic limb-threatening ischemia (CLTI) patients revascularisation surgery; for colorectal liver metastasis (CRLM) patients metastatic liver surgery
- Colorectal liver metastases (CRLM) group: All CRLM patients presenting with wound, ischemia, foot infection (WIfI) with stage IV disease consecutively treated at one institution
  Interventions: Procedure: For chronic limb-threatening ischemia (CLTI) patients revascularisation surgery; for colorectal liver metastasis (CRLM) patients metastatic liver surgery

INTERVENTIONS:
Procedure: For chronic limb-threatening ischemia (CLTI) patients revascularisation surgery; for colorectal liver metastasis (CRLM) patients metastatic liver surgery — For chronic limb-threatening ischemia (CLTI) patients that represents one of the revascularisation methods (endovascular, open surgery, hybrid).
  For the colorectal liver metastasis (CRLM) patients that represents liver resection with adjuvant chemo- or radiotherapy

SUMMARY:
Colorectal cancer (CRC) and chronic limb-threatening ischemia (CLTI) are relatively frequent and potentially fatal diseases. However, studies that are comparing clinical outcomes between CRC and CLTI patients in more advanced stages of the disease are lacking. The study aim was to evaluate outcomes of patients with colorectal cancer liver metastases (CRLM) treated by curative-intent liver resection and CLTI patients according to wound, ischemia, foot infection (WIfI) classification by comparing the short- and long-term clinical outcomes.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is characterized by a global pandemic of growing proportions. In 2016, The Global Burden of Disease study reported that 202 million adults worldwide have PAD, with a higher prevalence compared to ischaemic heart disease (154 million), Alzheimer's disease (64 million) and cancer (43 million). The patient prognosis after PAD occurrence is poor because the disease often progresses to chronic limb-threatening ischemia (CLTI) that is an end-stage disease.

The 5-year mortality risk in CLTI patients is about 60%. When the mortality risk of CLTI is compared to mortality rates of the most common malignant diseases only six of them have a higher 5-year mortality rate compared to CLTI. One of them is colorectal cancer (CRC). CRC is the third most commonly occurring cancer in men and the second most commonly occurring cancer in women.

According to the latest CLTI treatment guidelines, the Society for Vascular Surgery (SVS) WIfI (wound, infection, ischemia) classification should be employed to stage limb condition in patients with CLTI that is analog to the use of tumor, nodes, metastases (TNM) cancer staging system. Recent data indicate that WIfI appears to correlate strongly with important clinical outcomes.

The annual incidence of CLTI is greater than the incidence of cancers characterized by high mortality rates (esophageal, stomach, brain and ovarian). In addition, more people die from CLTI each year compared to death rates of the already mentioned cancers. However, studies that are comparing clinical outcomes between cancer and CLTI patients in more advanced stages of the disease are lacking.

The study aim was to evaluate outcomes of the wound, ischemia, foot infection (WIfI) stage IV CLTI and colorectal cancer liver metastases (CRLM) patients managed by curative-intent liver resection by comparing the short- and long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All chronic limb-threatening (CLTI) patients presenting with wound, ischemia, infection (WIfI) stage IV disease undergoing some revascularization procedure (endovascular, open surgery hybrid).
* All colorectal carcinoma (CRC) patients undergoing colorectal liver metastasis (CRLM) surgery

Exclusion Criteria:

* For CLTI group: patients who did not undergo revascularization surgery, those who underwent primary major amputation, patients with lower stages of the disease (stage I, II, and III), patients who had acute lower limb ischemia
* For the CRLM group we excluded patients who did not undergo curative surgery, those who underwent liver resection due to other malignancies (hepatocellular carcinoma, cholangiocarcinoma, etc.), patients who underwent palliative surgery, liver transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Chronic limb-threatening (CLTI)group - patients presenting with wound, ischemia, infection (WIfI) stage IV disease undergoing some revascularization procedure (endovascular, open surgery hybrid)
  * All colorectal carcinoma (CRC) patients undergoing colorectal liver metastasis (CRLM) curative surgery
Sampling Method: Non-Probability Sample
Enrollment: 836 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | up to 60 months
  Number of participants who died from all causes of death in both chronic limb-threatening ischemia (CLTI) and colorectal liver metastasis (CLRM) population in a given time period

SECONDARY OUTCOMES:
Short-term mortality | During the hospital stay (up to 30-days) and 30-day after the initial surgery
  Number of participants for both chronic limb-threatening ischemia (CLTI) and colorectal liver metastasis (CLRM) population who died in hospital, as well as 30 days after the initial surgery
Hospital adverse event | During the patients hospital stay (up to 30-days)
  Number of participants with the following postoperative adverse events: cardiac (acute coronary syndrome, heart failure, pulmonary embolism), pulmonary (intubation lasting longer than 72h, pneumonia, atelectasis requiring active treatment), hemodialysis, wound infection, postoperative surgical bleeding, red blood cell transfusion rate, hepatic insufficiency, biliary fistula, major amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Lazar Davidovic, MD PhD, Study Chair — Clinical Center of Serbia; Petar M Zlatanovic, MD, Principal Investigator — Clinical Center of Serbia
Locations (1):
- Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided
It will be made upon the reader's request